CLINICAL TRIAL: NCT04983589
Title: A Phase 3, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of BID Dosing of AGN-190584 in Subjects With Presbyopia
Brief Title: A Study to Assess Safety and Efficacy in Participants Age 40 to 55 With Presbyopia (Old Eye) Who Receive AGN-190584 in Both Eyes Twice Daily
Acronym: Virgo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M21-195
Record Dates: First submitted 2021-07-22; First posted 2021-07-30 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Presbyopia
Keywords: Presbyopia; AGN-190584; Pilocarpine HCl 1.25%; Old Eye; Aged Eye
MeSH Terms: conditions — Presbyopia | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vehicle (Placebo Comparator): Participants received vehicle, one drop bilaterally (in each eye), twice daily (BID), with a gap of 6 hours between both doses, for up to 14 days.
  Interventions: Drug: Vehicle
- AGN-190584 (Experimental): AGN-190584 ophthalmic solution, one drop bilaterally (in each eye), BID, with a gap of 6 hours between both doses, for up to 14 days.
  Interventions: Drug: Pilocarpine HCl

INTERVENTIONS:
Drug: Pilocarpine HCl — Pilocarpine HCl ophthalmic solution 1.25% ocular drops.
  Other Names: AGN-190584
  Arms: AGN-190584
Drug: Vehicle — Oxymetazoline HCl and pilocarpine HCl placebo ocular drops.
  Arms: Vehicle

SUMMARY:
Currently available treatments for presbyopia (old eye) include nonsurgical options (spectacles or contact lenses) and surgical options, however, each has its own risks and limitations. The purpose of this study is to evaluate how effective AGN-190584 is in treating presbyopia compared to vehicle (placebo).

AGN-190584 is an investigational drug being developed for the treatment of presbyopia. Participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to vehicle. Around 200 participants age 40-55 years with a diagnosis of presbyopia will be enrolled in the study in approximately 20 sites in the United States.

Participants will receive AGN-190584 or vehicle in each eye twice daily for 14 days.

There may be additional procedures for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a doctor's office. The effect of the treatment will be checked by medical assessments, vision/eye tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Objective and subjective evidence of presbyopia.

Exclusion Criteria:

* Corneal abnormalities (including keratoconus, corneal scar, Fuchs' endothelial dystrophy, guttata, or edema) in either eye that are likely to interfere with visual acuity.
* Narrow iridocorneal angles (Shaffer grade <=2 or lower on gonioscopy examination), history of angle-closure glaucoma, or previous iridotomy.
* Diagnosis of any type of glaucoma or ocular hypertension.
* History of cataract surgery, phakic intraocular lens surgery, corneal inlay surgery, radial keratotomy, or any intraocular surgery.
* Use of temporary or permanent punctal plugs or history of punctal cautery in one or both eyes.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (23):
- United States (23):
  - Empire Eye and Laser /ID# 231433, Bakersfield, California
  - Global Research Management /ID# 231300, Glendale, California
  - United Medical Research Institute /ID# 233982, Inglewood, California
  - North Valley Eye Medical Group, Inc. /ID# 231270, Mission Hills, California
  - The Eye Research Foundation /ID# 231274, Newport Beach, California
  - Martel Eye Medical Group /ID# 231332, Rancho Cordova, California
  - Nature Coast Clinical Research - Crystal River /ID# 231298, Crystal River, Florida
  - Bruce Segal, MD /ID# 231413, Delray Beach, Florida
  - Clayton Eye Clinical Research, LLC /ID# 231243, Morrow, Georgia
  - Jacksoneye, SC /ID# 231374, Lake Villa, Illinois
  - Price Vision Group /ID# 231261, Indianapolis, Indiana
  - Kannarr Eye Care /ID# 231363, Pittsburg, Kansas
  - Cincinnati Eye Institute- Edgewood /ID# 231356, Edgewood, Kentucky
  - The Eye Care Institute /ID# 231275, Louisville, Kentucky
  - Rochester Ophthalmological Group PC /ID# 231371, Rochester, New York
  - Southern College of Optometry /ID# 231325, Memphis, Tennessee
  - Total Eye Care, PA /ID# 231245, Memphis, Tennessee
  - Advancing Vision Research /ID# 231244, Smyrna, Tennessee
  - Hill Country Eye Center /ID# 231293, Cedar Park, Texas
  - The Cataract & Glaucoma Center /ID# 231292, El Paso, Texas
  - Eye associates /ID# 231262, San Antonio, Texas
  - Hoopes, Durrie, Rivera Research /ID# 231273, Draper, Utah
  - Country Hills Eye Center /ID# 231414, Ogden, Utah

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 22 investigational sites in the United States from 02 September 2021 to 11 February 2022.
Period: Overall Study
Arm/Group | Vehicle | AGN-190584
Started | 116 | 114
Completed | 113 | 111
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — COVID-19 Infection | 1 | 0
Not completed — COVID-19 Logistical Restrictions | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Vehicle: Participants received vehicle, one drop bilaterally (in each eye), BID, with a gap of 6 hours between both doses, for up to 14 days.
- Total: Total of all reporting groups
Arm/Group | Vehicle | AGN-190584 | Total
Number analyzed (Participants) | 116 | 114 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (3.87) | 50.4 (3.33) | 50.3 (3.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 70 | 132
  Male | 54 | 44 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 30 | 59
  Not Hispanic or Latino | 87 | 84 | 171
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 98 | 93 | 191
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-Contrast, Binocular Distance-Corrected Near Visual Acuity (DCNVA) With No More Than 5-Letter Loss in Mesopic Corrected Distance Visual Acuity (CDVA) With the Same Refractive Correction
Description: Visual acuity for near (40 centimeter [cm]) and distance (4 meter [m]) targets were measured in mesopic conditions using an eye chart. High contrast corrected distance visual acuity (CDVA) was assessed binocularly (in each eye) using the provided visual acuity charts for distance vision in a room with mesopic lighting conditions (10 to 11 lux) measured at the target. Both near vision and distance vision were measured to evaluate the effect of AGN-190584. A participant who gained 3 lines or more in mesopic, high contrast, binocular DCNVA with no more than 5-letter loss in mesopic CDVA with the same refractive correction was regarded as a responder. A participant with missing data was regarded as a non-responder.
Time Frame: 3 hours after second dose on Day 14
Population: ITT Population included all randomized participants. Percentages are rounded off to whole number at single decimal.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | AGN-190584
Number analyzed (Participants) | 116 | 114
percentage of participants | 7.8 | 35.1
Statistical Analysis 1: Comparison: Vehicle vs AGN-190584; Test type: Superiority; p < 0.0001, Chi-squared — Analysis was done using chi-square test; Percentage Difference = 27.3, 95% CI 2-sided [17.3 to 37.4] — The 95% confidence interval for the proportion differences was calculated using the normal approximation based on pooled variance without continuity correction

2. Secondary Outcome: Percentage of Participants Gaining 3 Lines or More in Photopic, High-Contrast, Binocular DCNVA With No More Than a 5-Letter Loss in Photopic CDVA With the Same Refractive Correction
Description: Visual acuity for near (40 centimeter [cm]) and distance (4 meter [m]) targets were measured in photopic conditions using an eye chart. High contrast corrected distance visual acuity (CDVA) was assessed binocularly (in each eye) using the provided visual acuity charts for distance vision in a room with photopic lighting conditions (≥ 251 lux) measured at the target. Both near vision and distance vision were measured to evaluate the effect of AGN-190584. A participant who gained 3 lines or more in photopic, high contrast, binocular DCNVA with no more than 5-letter loss in photopic CDVA with the same refractive correction was regarded as a responder. A participant with missing data was regarded as a non-responder.
Time Frame: 3 hours after second dose on Day 14
Population: ITT Population included all randomized participants. Percentages are rounded off to whole number at single decimal.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | AGN-190584
Number analyzed (Participants) | 116 | 114
percentage of participants | 6.0 | 32.5
Statistical Analysis 1: Comparison: Vehicle vs AGN-190584; Test type: Superiority; p < 0.0001, Chi-squared — Analysis was done using chi-square test; Percentage Difference = 26.4, 95% CI 2-sided [16.8 to 36.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Gaining 2 Lines or More in Mesopic, High-Contrast, Binocular DCNVA With No More Than a 5-Letter Loss in Mesopic CDVA With the Same Refractive Correction
Description: Visual acuity for near (40 centimeter [cm]) and distance (4 meter [m]) targets were measured in mesopic conditions using an eye chart. High contrast corrected distance visual acuity (CDVA) was assessed binocularly (in each eye) using the provided visual acuity charts for distance vision in a room with photopic lighting conditions (10 to 11 lux) measured at the target. Both near vision and distance vision were measured to evaluate the effect of AGN-190584. A participant who gained 2 lines or more in mesopic, high contrast, binocular DCNVA with no more than 5-letter loss in mesopic CDVA with the same refractive correction was regarded as a responder at that visit/timepoint. A participant with missing data was regarded as a non-responder.
Time Frame: 3 hours after second dose on Day 14
Population: ITT Population included all randomized participants. Percentages are rounded off to whole number at single decimal.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | AGN-190584
Number analyzed (Participants) | 116 | 114
percentage of participants | 25.9 | 60.5
Statistical Analysis 1: Comparison: Vehicle vs AGN-190584; Test type: Superiority; p < 0.0001, Chi-squared — Analysis was done using chi-square test; Percentage Difference = 34.7, 95% CI 2-sided [22.7 to 46.7] — The 95% confidence interval for the proportion differences was calculated based on the normal approximation using pooled variance without continuity correction

4. Secondary Outcome: Percentage of Participants Achieving 20/40 or Better in Mesopic, High-Contrast, Binocular DCNVA With No More Than a 5-Letter Loss in Mesopic CDVA With the Same Refractive Correction
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Both near vision and distance vision were measured to evaluate the effect of AGN-190584. A participant who achieved 20/40 or better in mesopic, high contrast, binocular DCNVA with no more than 5-letter loss in mesopic CDVA with the same refractive correction was regarded as a responder at that visit/timepoint. A participant with missing data was regarded as a non-responder.
Time Frame: 3 hours after second dose on Day 14
Population: ITT Population included all randomized participants. Percentages are rounded off to whole number at single decimal.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | AGN-190584
Number analyzed (Participants) | 116 | 114
percentage of participants | 24.1 | 44.7
Statistical Analysis 1: Comparison: Vehicle vs AGN-190584; Test type: Superiority; p = 0.001, Chi-squared — Analysis was done using chi-square test; Percentage Difference = 20.6, 95% CI 2-sided [8.6 to 32.6] — The 95% confidence interval for the proportion differences was calculated using the normal approximation using pooled variance without continuity correction

ADVERSE EVENTS:
Time Frame: SAEs and other AEs were collected from the time of study drug administration through study completion, an average of 15 days for each participant.
Description: Safety Population included all participants who received at least 1 administration of study treatment.
Arm/Group | Vehicle | AGN-190584
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/114
Other Adverse Events (participants affected / at risk) | 4/116 | 16/114
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=116) | AGN-190584 (N=114)
EYE IRRITATION (Eye disorders) | 0 (0) | 7 (16)
HEADACHE (Nervous system disorders) | 4 (4) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04983589/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT04983589/SAP_001.pdf